CLINICAL TRIAL: NCT02346578
Title: Multicenter, Prospective, Randomised and Comparative Study of AA Therapy and Early Administrating Enzalutamide in Participants With CRPC Previously Treated With CAB Therapy Using Bicalutamide.
Brief Title: Comparative Study of Alternative Antiandrogen (AA) Therapy and Early Initiating of Enzalutamide for Castration-resistant Prostate Cancer (CRPC) After Combined Androgen Blockade (CAB) Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taro Iguchi, MD, PHD (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Taro Iguchi, MD, PHD, Osaka City University Graduate School of Medicine, Osaka City University
Organization: Osaka City University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCUU-CRPC
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide; Flutamide

ARMS (2):
- Enzalutamide (Experimental): Enzalutamide 160 mg administered orally once a day as four 40-mg soft capsules
  Interventions: Drug: Enzalutamide
- Flutamide (Active Comparator): Flutamide 125 mg administered orally three times a day as one tablet after meal
  Interventions: Drug: Flutamide

INTERVENTIONS:
Drug: Enzalutamide
  Arms: Enzalutamide
Drug: Flutamide
  Arms: Flutamide

SUMMARY:
The objective of this study is to compare the efficacy and safety of enzalutamide or alternative AA therapy in CRPC participants who were previously treated with a combined androgen blockade therapy which included bicalutamide (Bic-CAB). Efficacy and safety of enzalutamide and alternative AA therapy will be evaluated, and effective therapy against CRPC after treatment with Bic-CAB will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone of less than 50 ng/dL
* Participants who was detected of disease progression on image or relapse of PSA (All PSA values measured 3 time at least one week interval are consecutively increased and final value is 2 ng/mL or more. If third value is not higher than second one, fourth measurement will be undertaken and its value must be higher than second one.)
* Participants who relapsed after CAB with bicalutamide
* Eastern Cooperative Oncology Group (ECOG) performance status is 0 or 1
* Aged 20 years or older
* Participants who provided written informed consent

Exclusion Criteria:

* Any prior treatment with enzalutamide, flutamide, abiraterone or chemotherapy, except for neoadjuvant therapy
* With active double cancer
* Any prior treatment with bicalutamide within 6 weeks
* Participants who received systemic biological therapy (except for existing approved drug for bone or treatment with luteinizing hormone-releasing hormone (LHRH) analogue) or received treatment with other antitumor agent for prostate cancer
* With serious complication
* History of hypersensitivity to enzalutamide or any other excipient of enzalutamide
* History of hypersensitivity to flutamide-containing agent
* With liver dysfunction
* Participants who are considered as inadequate by the investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-12; Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Percentage of participants whose prostate specific antigen (PSA) decreased 50 percent or more at month 3 | Month 3

SECONDARY OUTCOMES:
Percentage of participants whose PSA decreased 50 percent or more at month 6 | Month 6
Percentage of participants who showed disease progression at month 3 | Month 3
Percentage of participants who showed disease progression at month 6 | Month 6
PSA progression-free survival (PFS) | Up to 39 months
QOL measured by functional assessment of cancer therapy-prostate (FACT-P) | Up to 39 months

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka City University Graduate School of Medicine, Osaka, Japan

REFERENCES:
- [Background] Iguchi T, Tamada S, Kato M, Yasuda S, Yamasaki T, Nakatani T. Enzalutamide versus flutamide for castration-resistant prostate cancer after combined androgen blockade therapy with bicalutamide: study protocol for a multicenter randomized phase II trial (the OCUU-CRPC study). BMC Cancer. 2019 Apr 11;19(1):339. doi: 10.1186/s12885-019-5526-3. PMID 30971225
- [Result] Iguchi T, Tamada S, Kato M, Yasuda S, Machida Y, Ohmachi T, Ishii K, Iwata H, Yamamoto S, Kanamaru T, Morimoto K, Hase T, Tashiro K, Harimoto K, Deguchi T, Adachi T, Iwamoto K, Takegaki Y, Nakatani T. Enzalutamide versus flutamide for castration-resistant prostate cancer after combined androgen blockade therapy with bicalutamide: the OCUU-CRPC study. Int J Clin Oncol. 2020 Mar;25(3):486-494. doi: 10.1007/s10147-019-01554-3. Epub 2019 Sep 28. PMID 31564004